CLINICAL TRIAL: NCT03878069
Title: Single Arm, Open-Label, Multicenter, Registry Study of Revcovi (Elapegademase-lvlr) Treatment in ADA-SCID Patients Requiring Enzyme Replacement Therapy
Brief Title: Registry Study of Revcovi Treatment in Patients With ADA-SCID
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-06814AA1-01
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Adenosine Deaminase Severe Combined Immunodeficiency
Keywords: ADA-SCID; Revcovi; ERT
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency | interventions — elapegademase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with ADA-SCID in need of ERT treatment: All participants will receive Revcovi. For analysis purposes, there will be three groups, who differ with respect to ERT history:
  * Adagen-naïve: Subjects starting on ERT for the first time
  * Adagen-transitioning: Subjects switching from Adagen to Revcovi
  * STP-2279-002 participants: Subjects who had taken part in an earlier Phase III trial of Revcovi (study STP-2279-002) in which they had been switched from Adagen to Revcovi. This last group differs from the Adagen-transitioning group in that they will have been on Revcovi the longest.
  Interventions: Biological: elapegademase-lvlr

INTERVENTIONS:
Biological: elapegademase-lvlr — Revcovi is administered intramuscularly (i.m.). Weekly dosage is calculated in mg/kg of body weight, and can be adjusted over the course of the trial based on ADA activity and dAXP concentration as well as on clinical assessment by the treating physician.
  Other Names: Revcovi

SUMMARY:
This registry study is being conducted in patients with adenosine deaminase severe combined immune deficiency (ADA-SCID) who require enzyme replacement therapy (ERT) treatment with Revcovi. Data on safety and on measures of efficacy are collected.

DETAILED DESCRIPTION:
Patients with ADA-SCID who require ERT will receive Revcovi on a dosage and schedule determined by the treating physician. They will be followed for safety throughout the study, and will be monitored for the efficacy markers of adenosine deaminase (ADA) activity and deoxyadenosine nucleotide (dAXP) concentration according to a suggested schedule. Some subjects will be new to ERT; some will have transitioned from Adagen, which was the ERT available before Revcovi; and some will have previously participated in an earlier Phase 3 trial of Revcovi (study STP-2279-002). Patients will be followed either until they are able to successfully undergo a stem cell transplant or stem cell gene therapy and thus no longer require ERT treatment, or until all ongoing participants have received a minimum of 24 months of Revcovi treatment.

Note: Due to the nature of this study, all analyses are descriptive and no statistical hypotheses will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged newborn to adult
* In need of ERT treatment due to one of the following circumstances:

  * Waiting to receive a stem cell transplant
  * Previously declined, had been found to be ineligible for, or did not respond to a stem cell transplant
  * Waiting to enrol in a clinical trial on gene therapy, or had been found to be ineligible for or had failed such a trial
* One of the following histories of ERT treatment:

  * Revcovi only
  * Previously on Adagen but had transitioned to Revcovi
  * Not yet on any ERT but about to start on Revcovi

Exclusion Criteria:

* Any condition that, in the opinion of the Investigator, makes the patient unsuitable for the study.

Ages: 0 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ADA-SCID who require ERT
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of California Los Angeles, Los Angeles, California
  - Allergy & Asthma Medical Group and Research Center, A P.C., San Diego, California
  - UCSF - University of California, San Francisco, California
  - Children's National, Washington D.C., District of Columbia
  - University of South Florida Allergy Immunology Clinic, St. Petersburg, Florida
  - Childrens Hospital of New Orleans, New Orleans, Louisiana
  - Children's Minnesota, Minneapolis, Minnesota
  - St. Louis Children's Hospital - Washington University School of Medicine, St Louis, Missouri
  - UBMD Pediatrics Outpatient Center, Buffalo, New York
  - Duke University Hospital, Durham, North Carolina
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four of the participants had taken part in an earlier trial of Revcovi, study STP-2279-002, and were invited to continue in the registry study. The remaining participants were invited to enroll by their treating physicians.
Groups:
- Adagen-naive: Subjects starting on ERT for the first time
- Adagen-transitioning: Subjects switching from Adagen to Revcovi
- STP-2279-002 Participant: Subjects who had taken part in an earlier Phase III trial of Revcovi
Period: Overall Study
Arm/Group | Adagen-naive | Adagen-transitioning | STP-2279-002 Participant
Started | 7 | 21 | 4
Completed | 7 | 20 (One subject in the Adagen-transitioning group died during the study of causes unrelated to Revcovi treatment.) | 4
Not Completed | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adagen-naive | Adagen-transitioning | STP-2279-002 Participant | Total
Number analyzed (Participants) | 7 | 21 | 4 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 11 | 0 | 18
  Between 18 and 65 years | 0 | 10 | 4 | 14
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 15 | 2 | 20
  Male | 4 | 6 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 7
  Not Hispanic or Latino | 5 | 18 | 2 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 8 | 0 | 9
  White | 4 | 10 | 4 | 18
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 1
Number of subjects at or below the toxicity threshold for dAXP concentration [Count of Participants; unit: Participants] — A deficiency in the ADA enzyme results in a build-up of dAXP nucleotides (dAXP), which are toxic to lymphocytes and lead to impairment of immune function. A detoxified level of dAXP concentration is defined as a trough value of 0.02 millimoles per liter (mmol/L) or lower. Since the design of this study included some ADA-SCID patients who had been on an earlier enzyme replacement therapy (Adagen) prior to starting Revcovi and some who were starting it for the first time, it was of importance to see in both cases what the levels of dAXP were at baseline, prior to starting Revcovi.
  Participants | 0 | 13 | 4 | 17
Number of subjects meeting the optimal threshold for ADA activity [Count of Participants; unit: Participants] — An optimal level of ADA plasma activity is defined as a trough value of 30 millimoles per hour per liter (mmol/h/L) or above. Since the design of the study included some patients who had been on an earlier enzyme replacement therapy (Adagen) prior to starting Revcovi and some who were starting it for the first time, it was of importance to see in both cases what ADA levels were at baseline, prior to starting Revcovi.
  Note: For 6 of the naïve subjects, this measure was obtained after the start of Revcovi, so represents the early effects of treatment rather than actual pre-treatment status.
  Participants | 6 | 9 | 0 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Meeting the Toxicity Threshold for Deoxyadenosine Nucleotide (dAXP) Concentration at the Last Measurement
Description: A deficiency in the ADA enzyme results in a build-up of dAXP nucleotides, which are toxic to lymphocytes and lead to impairment of immune function. A detoxified level of dAXP concentration is defined as a trough value of 0.02 millimoles per liter (mmol/L) or lower. Data are presented as the number of subjects who met the targeted threshold at the final measurement, whether that took place at Month 24 or earlier.
Time Frame: From enrollment to end of treatment up to Month 24
Population: The As-Treated (AT) population, which included all subjects who received at least one dose of Revcovi.
Measure: Count of Participants; unit: Participants
Arm/Group | Adagen-naive | Adagen-transitioning | STP-2279-002 Participant
Number analyzed (Participants) | 7 | 21 | 4
Participants | 6 | 17 | 4

2. Primary Outcome: Number of Subjects Meeting the Optimal Threshold for ADA Activity at the Last Measurement
Description: An optimal level of ADA plasma activity is defined as a trough value of 30 millimoles per hour per liter (mmol/h/L) or greater. Data are presented as the number of subjects who met the targeted threshold at the final measurement, whether that took place at Month 24 or earlier.
Time Frame: From enrollment to end of treatment up to Month 24
Population: The As-Treated (AT) population, which included all subjects who received at least one dose of Revcovi.
Measure: Count of Participants; unit: Participants
Arm/Group | Adagen-naive | Adagen-transitioning | STP-2279-002 Participant
Number analyzed (Participants) | 7 | 21 | 4
Participants | 7 | 14 | 4

3. Primary Outcome: Safety of Revcovi
Description: The number of subjects reporting adverse events (AEs). Due to the nature of ADA-SCID, only AEs deemed to be at least possibly related to Revcovi treatment were documented.
Time Frame: From enrollment to end of treatment up to Month 24
Population: The As-Treated (AT) population, which included all subjects who received at least one dose of Revcovi.
Measure: Count of Participants; unit: Participants
Arm/Group | Adagen-naive | Adagen-transitioning | STP-2279-002 Participant
Number analyzed (Participants) | 7 | 21 | 4
Participants | 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: At any time during the study. Duration of participation was a minimum of 24 months, or until undergoing successful treatment with stem cell transplant or hematopoietic stem cell gene therapy.
Description: For mortality, all incidences are reported. For non-fatal serious adverse events (SAEs) and non-serious adverse events, due to the nature of the disease, sites were asked to report only those events deemed to be at least possibly related to Revcovi treatment, along with clinically meaningful laboratory abnormalities.
Groups:
- Patients With ADA-SCID in Need of ERT Treatment: All participants will receive Revcovi and will be monitored for adverse events (AEs) throughout their participation in the study. Only AEs deemed at least possibly related to Revcovi treatment will be documented.
Arm/Group | Patients With ADA-SCID in Need of ERT Treatment
All-Cause Mortality (participants affected / at risk) | 1/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 4/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With ADA-SCID in Need of ERT Treatment (N=32)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Exposure via skin contact (Injury, poisoning and procedural complications) | 1 (1)
Weight increased (Investigations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT03878069/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT03878069/SAP_001.pdf
  • Informed Consent Form (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT03878069/ICF_002.pdf